CLINICAL TRIAL: NCT01715597
Title: Placebo-controlled,Doubled,Randomized Trial Evaluating the Effect of Intravenous Ascorbic Acid on Intraoperative Blood Loss in Women Undergoing Laparoscopic Myomectomy
Brief Title: Study on the Effect of Intravenous Ascorbic Acid on Intraoperative Blood Loss in Women With Uterine Myoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Kidong Kim, Assistant professor in department of OBGY, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNUBH_GO_016
Record Dates: First submitted 2012-10-22; First posted 2012-10-29 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Uterine Leiomyoma
Keywords: uterine leiomyoma; laparoscopic myomectomy; intraoperative blood loss; ascorbic acid
MeSH Terms: conditions — Myofibroma | interventions — Ascorbic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ascorbic acid (Experimental): ascorbic acid 2g in normal saline 500ml IV start 2hours before the operation
  Interventions: Drug: ascorbic acid; Drug: Normal saline
- Control (Placebo Comparator): Normal saline 500ml IV infusion for 2hour
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: ascorbic acid — ascorbic acid 2g in normal saline 500ml IV start 30min before the operation and infusion for 2 hour
  Arms: ascorbic acid
Drug: Normal saline — normal saline 500ml IV

SUMMARY:
The investigators want to know whether the intravenous ascorbic acid would reduce the blood loss during laparoscopic myoma surgery. The investigators randomized patients into intravenous ascorbic acid group and placebo group and examined the blood loss in both groups.

ELIGIBILITY:
Inclusion Criteria:

* uterine myoma
* be planning to laparoscopic myomectomy
* images ; the number of myoma <4
* images ; the diameter of the largest myoma <9cm

Exclusion Criteria:

* be planning other surgery in addition to laparoscopy
* clinically significant coagulation abnormality

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-12; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
blood loss | during laparoscopic myomectomy

OTHER OUTCOMES:
time of operation | during laparoscopic myomectomy
the amount of transfusion | during laparoscopic myomectomy
the difference of hemoglobin | postoperative day 1
  postoperative day 1 hemoglobin - preoperative hemoglobin + hemoglobin increased by transfusion (hemoglobin 1 per RBC 1 pack transfusion)
acute urinary retention | 2days after the operation

CONTACTS AND LOCATIONS:
Overall Officials: kiding kim, M.D., Principal Investigator — Seoul National University Bundang Hospital,Gyeongg-ido,Republic of Korea
Locations (1):
- Seoul National University Bundang Hospital, Gyeongg-ido, South Korea

REFERENCES:
- [Derived] Lee B, Kim K, Cho HY, Yang EJ, Suh DH, No JH, Lee JR, Hwang JW, Do SH, Kim YB. Effect of intravenous ascorbic acid infusion on blood loss during laparoscopic myomectomy: a randomized, double-blind, placebo-controlled trial. Eur J Obstet Gynecol Reprod Biol. 2016 Apr;199:187-91. doi: 10.1016/j.ejogrb.2016.02.014. Epub 2016 Feb 21. PMID 26946313